CLINICAL TRIAL: NCT06424210
Title: The Role of Surgery for Esophageal Cancer With Metastatic Disease (M1)
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202211084RIND
Record Dates: First submitted 2024-05-13; First posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2023-02

CONDITIONS: Esophageal Cancer; Metastatic Disease
MeSH Terms: conditions — Esophageal Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Treatment of stage IV esophageal cancer is traditionally palliative, but treatment response is usually poor. The role of surgery in the treatment of advanced esophageal cancer remains controversial. We sought to determine whether surgical treatment followed by neoadjuvant chemoradiation therapy might provide survival benefits for these patients.

A retrospective review of esophageal cancer patients with M1 disease treated at National Taiwan University Hospital was performed from April 2002 to June 2021. Patient demographics and cancer staging, treatment, and disease recurrence, and time of follow up were included for analysis. Univariate and multivariate analysis was performed for overall survival and progression-free survival analysis. Propensity score matching based on patient age and tumor staging characteristics was also performed for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Stage IV Esophageal Cancer patients
* Patients were treated with chemoradiation therapy (CCRT)

Exclusion Criteria:

* Not Stage IV Esophageal Cancer patients
* Patients were not treated with chemoradiation therapy (CCRT)

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study enrolled a cohort of patients diagnosed with stage IV esophageal cancer who had tumor metastasis to distant organs, including lymph node metastasis detected in the retroperitoneum, which could not be eradicated by surgery, from April 2002 to June 2021 in a tertiary medical center.
Sampling Method: Non-Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Overall survival and progression-free survival | 5 years
  Overall survival (OS) and progression-free survival (PFS) curves of patients with or without esophagectomy in the entire study cohort of stage IV esophageal cancer with distant metastasis.

CONTACTS AND LOCATIONS:
Overall Officials: Jang-Ming Lee, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Zhongzheng, Taiwan